CLINICAL TRIAL: NCT05455112
Title: Phase IIb Clinical Trial to Evaluate the Efficacy and Safety of the Administration of RUTI® Immunotherapy With the Standard Treatment in Patients With Tuberculosis
Brief Title: Safety and Efficacy of RUTI® With the Standard of Treatment for Tuberculosis
Acronym: CONSTAN-ARG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Archivel Farma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONSTAN-ARG
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis, Pulmonary
Keywords: Tuberculosis, immunotherapy, drug-susceptible
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RUTI (Experimental): Single injection of RUTI 25µg of FCMtb at day 0.
  Interventions: Biological: RUTI® Vaccine
- Placebo (Placebo Comparator): Single injection of saline at day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RUTI® Vaccine — One subcutaneous injection of RUTI 25µg FCMtb
  Arms: RUTI
Biological: Placebo — One subcutaneous injection of saline
  Arms: Placebo

SUMMARY:
This study is proposed to evaluate the safety and efficacy of the RUTI vaccine in patients with pulmonary tuberculosis. Therapeutic vaccination of RUTI would stimulate the immune response not only against growing bacteria, but also against bacteria in a latent state that are less sensitive to antibiotic treatments. Therapeutic vaccination in patients with pulmonary tuberculosis could improve the speed of recovery of patients without inducing the appearance of drug resistance.

DETAILED DESCRIPTION:
The safety and immunogenicity of RUTI was established in healthy volunteers, patients with latent tuberculosis (TB); and Drug Susceptible (DS) -TB and Drug resistance (DR)-TB. This study proposed to evaluate the safety and efficacy of the RUTI vaccine in patients with active pulmonary TB. Immunotherapy for TB could shorten the sputum culture conversion, therefore reduce the time required to cure. Therapeutic vaccines do not interfere directly with the causative organism and hence, they are not involved in the development of drug resistance. Therapeutic vaccination would also be beneficial for DS-TB as it could increase the response to the standard therapy and help diminish the development of drug resistance. The vaccination stimulates the immune response during the continuation phase of TB treatment in which the remaining bacteria are poorly sensitive, if not refractory, to antimycobacterial agents, and potentiate chemotherapy. Reducing the huge reservoir of mycobacterium tuberculosis (DS or not) by vaccination strategies could ultimately accelerate elimination of the disease worldwide.

As per the results of the Phase II clinical trial in patients with latent TB, the best polyantigenic response was obtained with a dose of 25µg of RUTI vaccine and the second inoculation did not further increase the response. Based on these findings, a single dose of 25µg of vaccine will be used in the study.

The objective of this study is to i) explore the efficacy as reduction of bacillary load through the study of early bactericidal activity (EBA) in patients with DS-TB; and ii) provide data from safety perspective of the vaccine RUTI (25 µg FCMtb) in patients with TB, when given concomitant with the standard of care treatment initiation.

The study will include patients diagnosed with pulmonary DS-TB, candidate to start treatment with standard-care TB drugs and without any disease that could compromise the assessment of the response to the vaccination, or increase the risk of adverse events. RUTI will be administered on the day of TB treatment start, EBA will be measured on days 2, 4, 7, 10, 12, and 14, and adverse events will be collected up to week 24. Other measurements will be performed to assess the sputum culture conversion (SCC), clinical, X-ray or laboratory worsening, improvement of clinical signs and symptoms, and health-related quality-of-life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older
* Written informed consent
* Laboratory confirmed pulmonary TB
* Clinical symptoms compatible with pulmonary TB and/or X-ray evidence of pulmonary TB
* Women of non-childbearing potential: at least 2 years post-menopausal or surgically sterile (e.g. tubal ligation)
* Women of childbearing potential (including women less than 2 years past menopause) must have a negative pregnancy test at enrollment and must agree to use dual-barrier methods of contraception, intrauterine device (IUD), bilateral tubal occlusion, sexual abstinence, or vasectomized partner.
* Males must agree to use a double barrier method of contraception at least 1 month after RUTI/placebo vaccination; or the male patient or his female partner must be surgically sterile or the female partner must be post-menopausal
* Willing and able to attend all study visits and comply with all study procedures
* Verifiable address or place of residence easy accessible to perform visits and willing to inform the research team of any change during the treatment and follow-up period

Exclusion Criteria:

* Unable to provide written informed consent
* Women reported, or detected, or willing to be pregnant during the trial period; Men willing to conceive a child during the study or 6 months after end of treatment
* Severity of illness precluding full evaluation: expected early death, evidenced by respiratory failure, low blood pressure, WHO performance score 3-4
* Evidence or suspicion of resistance to rifampin, isoniazid, pyrazinamide, and ethambutol, either laboratory-confirmed or based on epidemiological history at screening
* Previous treatment for M. tuberculosis in the previous 24 months.
* Bodyweight < 40kg
* Unstable Diabetes Mellitus as a poor metabolic control within the past 12 months
* HIV-infected subjects
* Major co-morbid conditions or any other finding which in the opinion of the investigator would compromise the protocol compliance or significantly influence the interpretation of results
* HIstory of severe mental ilness which, in the opinion of the investigator, may exclude the participant from participating in the trial.
* Any of the following laboratory parameters:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN)
  * Total bilirubin > 2 x ULN
  * Neutrophil count ≤ 500 neutrophils / mm3
  * Platelet count < 50,000 platelets / mm3
* Alcohol use: potential participant either self-reports or in the investigator's opinion that the patient drinks more than an average of four units/day over a usual week or is a binge drinker (men: 5 or more drinks; women: consume 4 or more drinks, in about 2 hours)
* Known allergy or any hipersensitivity to study mediactions, including rifampin, isoniazid, pyrazinamide, and ethambutol, or any of its excipients.
* Documented allergy to anti-TB vaccines or any excipient of the RUTI vaccine.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Early bactericidal activity (EBA) 0-14 | From day 0 to day 14
  Change in EBA, using the time to positivity (TTP) of sputum in liquid Mycobacteria Growth Indicator Tube (MGIT)
Adverse events | From day 0 to week 24
  Proportion of patients with treatment-emergent adverse events (TEAE)
Grade 3-4 adverse events | From day 0 to week 24
  Total number of grade 3 and 4 adverse events (AE)

SECONDARY OUTCOMES:
Time to sputum culture conversion (SCC) | From day 0 to week 16
  Time to SCC, in liquid MGIT
Proportion of SCC at week 16 | From day 0 to week 16
  Proportion of participants with SCC, in liquid MGIT
Proportion of SCC at week 16 | From day 0 to week 8
  Proportion of participants with SCC, in liquid MGIT
Early bactericidal activity (EBA) 2-14 | From day 2 to day 14
  Change in EBA, using the TTP of sputum in liquid MGIT
Early bactericidal activity (EBA) 7-14 | From day 7 to day 14
  Change in EBA, using the TTP of sputum in liquid MGIT
Early bactericidal activity (EBA) 24 weeks | From day 0 to week 24
  Change in EBA, using the TTP of sputum in liquid MGIT
Proportion of SCC per weeks | Weeks 4, 12, 16, and 24
  Proportion of participants with SCC, in liquid MGIT
Clinical worsening | From day 0 to week 24
  Proportion of participants with clinical, X-ray, or laboratory worsening
Improvement of clinical signs and symptoms | Weeks 1, 2, 8, 12, 16, and 24.
  Proportion of participants with improvement on Bandim TB score
Improvement of quality of life | Weeks 8 and 24
  Proportion of participants with improvement on health-related quality of life (HRQOL)
Discontinuation of TB treatment | From day 0 to week 24.
  Proportion of participants who discontinue treatment due to failure, resistance, other.

CONTACTS AND LOCATIONS:
Locations (2):
- Argentina (2):
  - Hospital José Nestor Lencinas, Godoy Cruz, Mendoza Province
  - Hospital de Clínicas Presidente Dr. Nicolás Avellaneda, San Miguel de Tucumán, Tucumán Province